CLINICAL TRIAL: NCT00725673
Title: Determination of Risk Factors for Developing Osteoporosis in COPD GOLD II Patients. A Case Control Study to Identify Possible Risk Factors for Developing Osteoporosis in COPD GOLD II Patients.
Brief Title: Case Control Study: Determinants of Osteoporosis in GOLD II COPD Patients.
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: L. Graat-Verboom/drs, Catharina Hospital Eindhoven
Other Study IDs: M07-1752; 18223
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Osteoporosis
Keywords: COPD; Osteoporosis; BMD; DEXA-scan
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: GOLD II COPD patients with osteoporosis
- 2: GOLD II COPD patients with a normal bone mineral density

SUMMARY:
Patients with COPD have been found to have an increased risk of osteoporosis. The underlying mechanism is not clear yet. This case control study aims to identify risk factors for osteoporosis in GOLD II COPD patients. COPD GOLD II patients with osteoporosis (cases) will be matched by gender and age to COPD GOLD II patients without osteoporosis(controls).

Possible risk factors for osteoporosis are:

* BMI/VVMI (body composition)
* emphysema vs chronic bronchitis
* physical capacity
* Use of certain medication (eg corticosteroids, SSRI's)
* Nutritional status
* Infectious parameters Outpatients from the pulmonary ward of the Catharina Hospital Eindhoven with GOLD II COPD according to the ATS and GOLD-guidelines will be included in the study (after written informed consent).

A DEXA-scan will be made, if patients are osteoporotic or have a normal BMD they will be included in the study.

A HRCT will be made, a six minutes walking distance will be performed, blood will be drawn for lab. analysis, an X-ray of the vertebral collum will be made, impedance will be measured and hight and weight will be measuered. Also patients will fill in a questionaire.

By univariate and multivariate analysis the collected data will be analysed to determine possible risk factors for th development of osteoporosis in COPD GOLD II patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 40 years
* GOLD II COPD
* Written permission

Exclusion Criteria:

* Age < 40 years
* No COPD or COPD GOLD I, III or IV
* no written permission

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GOLD II COPD patients (ATS and GOLD guidelines) visiting the outpatient clinic of pulmonary medicine of the Catharina Hospital Eindhoven.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Risk factors for osteoporosis in GOLD II COPD patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lidwien Graat-Verboom, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, North Brabant, Netherlands